CLINICAL TRIAL: NCT03327337
Title: Arthroscopic Assisted Balloon Tibioplasty for the Treatment of Schatzker II-IV Tibial Plateau Fractures
Acronym: AABTFTPF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2017-08-105
Record Dates: First submitted 2017-09-18; First posted 2017-10-31 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Arthroscopy; Tibial Fractures; Orthopedic; Fracture Fixation
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): operate with Arthroscopic Assisted Balloon Tibioplasty on this group patients
  Interventions: Procedure: Arthroscopic Assisted Balloon Tibioplasty
- control group (Other): operate with open reduction and internal fixation on this group patients
  Interventions: Procedure: Arthroscopic Assisted Balloon Tibioplasty

INTERVENTIONS:
Procedure: Arthroscopic Assisted Balloon Tibioplasty — Under arthroscopy, the balloon supports the articular surface, with additional bone graft and necessary internal fixation

SUMMARY:
The investigators use existing resources to carry out this new technology, in accord with the standard of the patients, were randomized to traditional fracture balloon tibia fixation or arthroscopic reduction under angioplasty, the original data and data acquisition in a certain period of time corresponding to the patient, through statistical and epidemiological analysis and comparison of the method of professional data analysis discussion and experience according to the analysis results, the balloon angioplasty tibial arthroscopy and traditional open reduction and internal fixation for the clinical differences between postoperative recovery of tibial plateau articular surface reduction and joint function, and feedback the results to guide the clinical diagnosis and treatment.

DETAILED DESCRIPTION:
The Balloon Tibioplasty arthroscopic assisted forming technique based on the existing data, the subject of the design, 1. patients met the inclusion criteria, were randomized to traditional fracture tibial fixation or balloon assisted arthroscopic reduction under angioplasty, through follow-up, statistical evaluation after operation were compared between the two techniques for clinical curative effect the difference of tibial plateau articular surface reduction and recovery of joint function. 2., through the clinical practice, operation and experience summary, found that the new technology in the operation of the existing deficiencies, in order to improve the technology. 3 guide clinical diagnosis and treatment through results feedback and analysis.The investigators use existing resources to carry out this new technology, in accord with the standard of the patients, were randomized to traditional fracture balloon tibia fixation or arthroscopic reduction under angioplasty, the original data and data acquisition in a certain period of time corresponding to the patient, through statistical and epidemiological analysis and comparison of the method of professional data analysis discussion and experience according to the analysis results, the balloon angioplasty tibial arthroscopy and traditional open reduction and internal fixation for the clinical differences between postoperative recovery of tibial plateau articular surface reduction and joint function, and feedback the results to guide the clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* fresh closed fracture X-ray and CT examination confirmed Schatzker II-IV type tibial plateau fracture patients.
* the patient signed the informed consent.

Exclusion Criteria:

* Pathologic fractures, patients with neurologic disorders, and skeletally immature patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rasmussen scores change after surgery | 3、6、12 and 24 mouth Rasmussen scores change after surgery
  the knee joint Rasmussen scores change after surgery
Rasmunssen radiological evaluation scores change after surgery | immediately, and at 2 weeks and 1, 3, 6, 12, and 24 months Rasmunssen radiological evaluation scores change after surgery
  Rasmunssen radiological evaluation scores change after surgery
The quality of reduction | 2 weeks and 1, 3, 6, 12, and 24 months postoperatively.
  The quality of reduction will be determined based on postoperative CT scans, which can directly measure the amount of residual depression

SECONDARY OUTCOMES:
Intraoperative blood loss | Operation day
  blood loss in surgery
Surgical duration | The day of the operation
  Surgical duration
VAS pain scores change after surgery | from the day of the operation to the day of discharge from hospital (up to 2 weeks).
  The severity of lower limb pain after surgery
Hospitalization period after surgery | The day of the operation to the day of discharge
  Hospitalization period after surgery
Complications | 1, 3, 6, 12, and 24 months follow-up time. (PTA may not be seen in patients within the 24-month follow-up period, and we will perform follow-up for at least 10 years in all patients.)
  Complications including wound infection, reoperations, and posttraumatic arthritis (PTA) will be recorded.
the Short-Form Health Survey (SF-36) questionnaire | 1, 3, 6, 12, and 24 months follow-up time
  Health-related quality of life will be measured using the Short-Form Health Survey (SF-36) questionnaire during follow-up.

REFERENCES:
- [Derived] Wang JQ, Jiang BJ, Guo WJ, Zhang WJ, Li AB, Zhao YM. Arthroscopic-assisted balloon tibioplasty versus open reduction internal fixation (ORIF) for treatment of Schatzker II-IV tibial plateau fractures: study protocol of a randomised controlled trial. BMJ Open. 2018 Aug 8;8(8):e021667. doi: 10.1136/bmjopen-2018-021667. PMID 30093519

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT03327337/Prot_SAP_000.pdf